CLINICAL TRIAL: NCT03520140
Title: Prevalence of Familial Hypercholesterolaemia (FH) in Italian Patients With Coronary Artery Disease
Acronym: POSTER
Status: Completed | Type: Observational
Sponsor: Heart Care Foundation (Other)
Collaborators: Fondazione SISA (Unknown)
Responsible Party: Sponsor
Other Study IDs: K18
Record Dates: First submitted 2018-04-13; First posted 2018-05-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease
Keywords: Familial hypercholesterolemia; Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Full gene sequencing of the genes involved in FH (LDLR, APOB, PVSK9 and LDLRAP1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the prevalence of familial hypercholesterolemia (FH) in patients with documented coronary artery disease (CAD) event [acute myocardial infarction (AMI), acute coronary syndrome (ACS), coronary artery bypass graft (CABG) or percutaneous coronary intervention (PCI)] followed by 100 cardiological centers representative of the whole Italian territory

DETAILED DESCRIPTION:
Familial hypercholesterolemia (FH) is a disease that causes exposure to elevated plasma levels of LDL cholesterol (LDL-C, low-density lipoprotein) and increasing the risk of premature coronary heart disease (coronary artery disease, CAD). The FH is a co-dominant genetic disease and can occur in heterozygous and homozygous form, with different severity. The prevalence in whites is estimated to be 1.500 for heterozygous familial hypercholesterolemia (HeFH) and 1.1000000 for homozygous familial hypercholesterolemia (HoFH). This prevalence is probably an underestimate, as it is based on prevalence rates in in-patient and disease registries, and is influenced by the early mortality of patients with FH. The situation does not improve if we consider patients admitted for acute coronary event (myocardial infarction - AMI and / or unstable angina, - ACS). If we consider LDL cholesterol cumulative load in a person affected by FH, the best approach intervention to reduce cardiovascular mortality is an early diagnosis and treatment.

The primary aim of the study is to evaluate the prevalence of FH in patients with documented CAD event (AMI, ACS, CABG or PCI) followed by 100 cardiologic centers representative of the whole Italian territory. The results will also permit to increase the cardiologists awareness of FH. Secondary objective will be the validation of Dutch Lipid Clinic Network (DLCN) criteria (annex 1), in the Italian CAD population (12). The characterization of the patients, carried out during the study, will allow to identify the priorities for health inteventions aimed at improving the FH diagnosis in the general population through the a cascade screening in the relatives of the genetically characterized subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a documented coronary artery disease, more precisely:

ACS PCI CABG The index event must be occurred between 15 days and 8 weeks preceding the enrollment.

- Written informed consent to participate to the study

Exclusion Criteria:

* Patients unwilling to give their written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have a documented coronary artery disease, more precisely:
  ACS PCI CABG The index event must be occurred between 15 days and 8 weeks preceding the enrollment
Sampling Method: Probability Sample
Enrollment: 5415 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Familial hypercholesterolemia diagnosis | Inclusion
  Dutch Lipid Clinic Network Score (DLCNS) for FH The DLCNS is a validated set of criteria based on the patients family history of premature cardiovascular disease (CVD) in their first degree relatives, their own CVD history, their untreated lipid levels and physical signs such as the presence of tendon xanthomata or arcus cornealis prior to the age of 45. The subsequent score categorizes patients by the likelihood of Familial Hypercholesterolaemia (FH) diagnosis.
  Definite FH if score >8 Probable FH if score 6-8 Possible FH if score 3-5 Unlikely FH if score <3
Genetic examination | Inclusion
  Sequencing of (LDLR, APOB, PVSK9 and LDLRAP1)

CONTACTS AND LOCATIONS:
Locations (81):
- Italy (81):
  - Istituto Scientifico Inrca - Uo Cardiologia/Utic/Telecardiologia, Ancona
  - Ospedali Riuniti - Sod Cardiologia Ospedaliera Emod. E Utic, Ancona
  - Osp. Andria Canosa - Po Andria - Cardiologia - Utic, Andria
  - Ospedale Generale Regionale-Po U. Parini - U.O. Cardiologia E Cure Intensive Card., Aosta
  - Ospedale Civile - U.O.C. Cardiologia, Arzignano
  - Ospedale Gen.Le Prov.Le C.G. Mazzoni - Sc Cardiologia, Ascoli Piceno
  - Ospedale E. Muscatello - U.O. Di Cardiologia - Utic, Augusta
  - Presidio Ospedaliero Moscati - U.O.C. Cardiologia, Aversa
  - Ospedale Policlinico - U.O. Cardiologia Universitaria, Bari
  - Ospedale San Paolo - Cardiologia-Utic, Bari
  - Azienda Ospedaliera G. Rummo - Cardiologia Interventistica E Utic, Benevento
  - Ospedale Maggiore - U.O. Di Cardiologia, Bologna
  - Ospedale Generale Regionale - Ospedale Generale Regionale Divisione Di Cardiologia, Bolzano
  - Ospedale Ss. Trinita' - S.C. Di Cardiologia, Borgomanero
  - Azienda Ospedaliera G. Brotzu - Struttura Complessa Di Cardiologia, Cagliari
  - Ospedale San Giovanni Di Dio - Clinica Cardiologica, Cagliari
  - Ospedale A. Cardarelli - U.O. Cardiologia E Utic, Campobasso
  - Presidio Ospedaliero F. Ferrari - Cardiologia - Utic, Casarano
  - Az. Ospedaliera S. Anna E S. Sebastiano - U.O. Cardiologia-Utic, Caserta
  - P.O. Garibaldi-Nesima - U.O.C. Di Cardiologia, Catania
  - Fondazione G. Giglio - U.O. Cardiologia E Utic, Cefalù
  - Ospedale Bassini - U.O. Cardiologia E Utic, Cinisello Balsamo
  - Ospedale Di Cittadella - U.O. Cardiologia, Cittadella
  - Ospedale San Giuseppe Da Copertino - U.O. Di Cardiologia-Utic, Copertino
  - Ospedale Valdichiana Santa Margherita - Uos Cardiologia E Hdu, Cortona
  - Maria Cecilia Hospital - U.O. Di Cardiologia, Cotignola
  - Ospedale Di Cremona - Uo Di Cardiologia, Cremona
  - Ospedale Civile Sant'Antonio Abate - U.O.C. Di Cardiologia E Utic, Erice
  - Ospedale Civile - U.O.C. Cardiologia - Utic, Fidenza
  - Aou Careggi - Interventistica Cardiologica Strutturale, Florence
  - Aou Careggi - Riabilitazione Cardiologica, Florence
  - Ospedale Santa Maria Nuova - Hdu Cardiologica/Utic, Florence
  - Ospedali Riuniti - S.C. Di Cardiologia Univ.-Utic, Foggia
  - Ospedale G.B. Morgagni - L. Pierantoni - U.O. Cardiologia, Forlì
  - E.O. Ospedali Galliera - S. C. Cardiologia, Genova
  - Ospedale Civile - Sc Cardiologia Area Nord, Guastalla
  - Citta' Di Lecce Hospital - U.O. Di Cardiologia, Lecce
  - Nuovo Ospedale Versilia - Sc Cardiologia, Lido di Camaiore
  - Ospedale Civile M. Giannuzzi - Cardiologia E Utic, Manduria
  - Presidio Ospedaliero Paolo Borsellino - U.O.C Cardiologia- Utic, Marsala
  - Ospedale G. Fucito - U.O. Di Cardiologia E Utic, Mercato San Severino
  - Policlinico Di Monza - Uo Cardiol. Clinica E Scompenso Cardiaco, Monza
  - Aorn Cardarelli - U.O. Cardiologia Con Utic, Napoli
  - Aorn Osp. Dei Colli- Po Vincenzo Monaldi - U.O.C. Cardiologia - S.U.N., Napoli
  - Aou Maggiore Della Carita' - Cardiologia Ii, Novara
  - Ospedale San Francesco - Cardiologia - Utic, Nuoro
  - Ospedale San Luigi Gonzaga - S.C.D.O. Cardiologia, Orbassano
  - Maria Eleonora Hospital - Cardiologia, Palermo
  - Ospedale Civico - U.O. Cardiologia, Partinico
  - Centro Cuore Morgagni - U.F. Utic Ed Emodinamica, Pedara
  - Ospedale Civile Ave Gratia Plena - U.O. Di Cardiologia E Utic, Piedimonte Matese
  - Ospedale San Jacopo - U.O. Cardiologia, Pistoia
  - Policlinico Citta' Di Pomezia S. Anna - U.O. Cardiologia-Utic, Pomezia
  - Ospedale Santa Maria Delle Grazie - U.O. Cardiologia - Utic, Pozzuoli
  - Arcispedale Santa Maria Nuova - S.C. Cardiologia, Reggio Emilia
  - Ospedale Infermi - U.O. Cardiologia, Rimini
  - Campus Biomedico - Cardiologia, Roma
  - Ospedale Madre Giuseppina Vannini - U.O.C. Cardiologia, Roma
  - P.O. San Filippo Neri - Asl Roma 1 - Uoc Cardiologia E Utic, Roma
  - Policlinico Casilino - U.O. Cardiologia, Roma
  - Policlinico Umberto Primo - Cardiologia B - Cardiologia E Angiologia, Roma
  - A.O.U.S. Giovanni Di Dio-Ruggi D'Aragona - Sc Di Cardiologia, Salerno
  - Ospedale G. Fracastoro - U.O.C. Di Cardiologia, San Bonifacio
  - Ospedale Casa Sollievo Della Sofferenza - Cardiologia - Utic - Riabil Cardiologica, San Giovanni Rotondo
  - Presidio Ospedaliero - U.O. Cardiologia, Sanremo
  - Ospedale San Giuseppe E Melorio - U.O.C. Cardiologia Utic, Santa Maria Capua Vetere
  - Presidio Ospedaliero Di Saronno - U.O.C. Di Cardiologia, Saronno
  - Ospedale Ignazio Veris Delli Ponti - Uoc Cardiologia-Utic, Scorrano
  - IRCCS Policlinico Multimedica - UO Cardiologia, Sesto San Giovanni
  - Ospedale San Matteo Degli Infermi - Servizio Di Cardiologia Con Utic, Spoleto
  - Ospedale Umberto I - Uoc Cardiologia E Utic, Syracuse
  - Casa Di Cura Villa Verde - Cardiologia, Taranto
  - Ospedale San Timoteo - Ssd Cardiologia Emodinamica, Termoli
  - Centro Polifunzionale Boldrini - Cardiologia Riabilitativa-Cardioaction, Thiene
  - Aou Citta' Della Salute E Della Scienza-Scdu Cardiologia, Torino
  - Ospedali Treviglio-Caravaggio - Cardiologia, Treviglio
  - Ospedali Riuniti - Osp. Maggiore - A.F. Cardiologia E Riabilitazione Cardio, Trieste
  - Pou Santa Maria Della Misericordia - S.O.C. Cardiologia, Udine
  - Ospedale Di Circolo E Fondazione Macchi - Ssd Unita' Di Cure Intensive Coronariche, Varese
  - Ospedale San Pio Da Pietrelcina - Cardiologia, Vasto
  - Ics Maugeri Spa Societa' Benefit - Uo Cardiologia Riabilitativa, Veruno

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gulizia MM, Maggioni AP, Abrignani MG, Bilato C, Mangiacapra F, Sanchez FA, Piovaccari G, Montagna L, Marini M, De Biasio M, Averna M, Casula M, Colivicchi F, Fabbri G, Lucci D, Zampoleri V, Catapano AL; POSTER Investigators. Prevalence Of familial hypercholeSTerolaemia (FH) in Italian Patients with coronary artERy disease: The POSTER study. Atherosclerosis. 2020 Sep;308:32-38. doi: 10.1016/j.atherosclerosis.2020.07.007. Epub 2020 Jul 29. PMID 32823190
- [Derived] Qureshi N, Da Silva MLR, Abdul-Hamid H, Weng SF, Kai J, Leonardi-Bee J. Strategies for screening for familial hypercholesterolaemia in primary care and other community settings. Cochrane Database Syst Rev. 2021 Oct 7;10(10):CD012985. doi: 10.1002/14651858.CD012985.pub2. PMID 34617591